CLINICAL TRIAL: NCT01051739
Title: Improved Assessment of Visual Field Change
Brief Title: Variability in Perimetry Study
Acronym: VIPII
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C7098-R
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma
Keywords: vision testing; perimetry; glaucoma; test variability
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: glaucoma
  Interventions: Procedure: Comparison of four visual field testing strategies
- Group 2: normal
  Interventions: Procedure: Comparison of four visual field testing strategies

INTERVENTIONS:
Procedure: Comparison of four visual field testing strategies — We compared the ability of four perimetric strategies to detect visual field change in the glaucoma arm.

SUMMARY:
Improved Assessment of Visual Field Change is a trial aimed at investigating mechanisms of visual field testing variability. The investigators have found using larger stimulus size substantially lowers short-term variability. In this study, the investigators will determine if larger stimuli detect visual field change at an earlier time. The investigators are also developing a statistical model that accounts for correlations of neighboring test locations.

DETAILED DESCRIPTION:
Disease of the optic nerve, including glaucoma, is the leading cause of blindness in the United States. Treatment decisions for optic nerve diseases are based largely on the changes in visual function that occur mostly as a consequence of disease progression. Unfortunately, the decision as to whether change of visual function has occurred is often difficult because of the high retest variability of conventional visual field testing (perimetry). This variability is so high that with moderate visual loss, a minimum of six tests are often needed in patients with optic nerve damage to reliably distinguish visual field deterioration from random variation. The preliminary data show that a substantial portion of the variability of perimetry lies in the type of stimulus used and the testing strategy applied.

OBJECTIVES: The investigators propose to test the hypothesis that a large portion of total perimetric variability in patients with visual loss is due to a poor signal-to-noise ratio associated with using a small fixed-size stimulus.

RESEARCH PLAN AND METHODS: To test this hypothesis, the investigators are examining patients with optic nerve diseases with conventional automated perimetry (size III) and tests having large-sized and scaled stimuli (size V, size VI (custom perimeter) and luminance size threshold perimetry - a test where threshold is found by changing stimulus size rather than stimulus intensity). Over four years the investigators will test 100 patients with and glaucoma and 60 normals each eight times. In addition, the investigators are retesting 50 subjects once a week for 5 weeks. The investigators are also studying the associated structural-functional correlations using OCT and developing a statistical model that accounts for correlations of neighboring test locations.

Perimetric variability and the reliable identification of visual field change is the single most difficult problem in visual testing today. The investigators anticipate identifying a method that allows efficient and accurate determination of visual field change. Identification of a superior method would (1) reduce the number of examinations needed, thereby reducing the costs of medical care; (2) minimize misdiagnosis, unnecessary testing and even unnecessary surgery that results from mistakenly interpreting fluctuation of the visual field as progression or improvement; (3) allow earlier disease intervention and (4) reduce the costs of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Mean deviation of -20 or better with 5-8 points (optimally 10 points) with a value of p= 0.05 or better on the total deviation plot
* Mild cataract with VA of 20/30 or better pinholed
* Refractive error of = to or less than 6 diopters with = or less than 3.50 diopters of cylinder
* Pupil diameter of 3 mm minimum
* Controlled hypertension, diabetes, migraine
* Pseudophakic/refractive surgery if no vision problems
* Trabeculectomy okay

Exclusion Criteria:

* History of other ocular or neurologic disease or surgery
* History of stroke
* Systemic disease [lupus, graves, cancer (within the last 5 yrs), AIDS, other]
* History of amblyopia
* Unreliable patient
* Frequently misses appointments
* Tests poorly
* Ocular hypertension
* Retinal problems
* Diabetic retinopathy
* Neurological disease (IIH, ON, AION)
* Cancer not in remission for the last 5 years
* Vein or artery occlusions
* Macular degeneration
* Trauma with vision loss
* Ocular inflammation (pars planitis, iritis, temporal aeuritis)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma patient with 0 to -25 dB mean deviation and normal subjects
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wall, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wall M, Doyle CK, Eden T, Zamba KD, Johnson CA. Size threshold perimetry performs as well as conventional automated perimetry with stimulus sizes III, V, and VI for glaucomatous loss. Invest Ophthalmol Vis Sci. 2013 Jun 7;54(6):3975-83. doi: 10.1167/iovs.12-11300. PMID 23633660
- [Background] Kummet CM, Zamba KD, Doyle CK, Johnson CA, Wall M. Refinement of pointwise linear regression criteria for determining glaucoma progression. Invest Ophthalmol Vis Sci. 2013 Sep 19;54(9):6234-41. doi: 10.1167/iovs.13-11680. PMID 23908183
- [Result] Wall M, Doyle CK, Zamba KD, Artes P, Johnson CA. The repeatability of mean defect with size III and size V standard automated perimetry. Invest Ophthalmol Vis Sci. 2013 Feb 15;54(2):1345-51. doi: 10.1167/iovs.12-10299. PMID 23341012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We completed recruitment in the first three years of the grant period at out Visual Field Laboratory at the University of Iowa
Pre-assignment Details: see inclusion and exclusion criteria
Groups:
- Group 1: glaucoma patients
- Group 2: normal ocular healthy controls
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 120 | 60
Completed | 92 | 47
Not Completed | 28 | 13
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 25 | 10

BASELINE CHARACTERISTICS:
Groups:
- Group 1: glaucoma with mean deviation from 0 to -25 dB
- Group 2: normal - healthy observers with no eye pathology other than refractive error less than 6 diopters of correction.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 41 | 66
  >=65 years | 95 | 19 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 61 (9) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 43 | 116
  Male | 47 | 17 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Progressing in Each Group Using Pointwise Linear Regression
Description: Perimetric method that most efficiently detects visual field change. secondary outcome: number of subjects progressing in each group using pointwise linear regression Linear regression was used to determine visual field worsening (progression) at each of 52 test locations. We required 3 or more worsening test locations at a p = 0.05 significance level for their to be significant progression.
Time Frame: 4 years
Population: Those that completed study
Measure: Number; unit: participants
Groups:
- Glaucoma: mean deviation 0 to -25 dB
- Control: Age-matched healthy observers were tested at baseline and then every six months for 4 years
Arm/Group | Glaucoma | Control
Number analyzed (Participants) | 92 | 47
participants | 0 | 0
Statistical Analysis 1: Comparison: Glaucoma vs Control; Test type: Superiority or Other; p = .21, Kaplan Meyer survival curves — The a priori threshold of statistical significance is p<0.05

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/60
Other Adverse Events (participants affected / at risk) | 0/120 | 0/60

LIMITATIONS AND CAVEATS:
not all subjects completed the study (dropouts).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes